CLINICAL TRIAL: NCT05409443
Title: Conventional or Bipolar Radiofrequency Ablation for the Treatment of Sacroiliac Joint Pain? The COBRA-SIJ Study, a Double-blinded, Randomized, Comparative Trial.
Brief Title: Conventional vs Bipolar SIJ RFA for Treatment of Sacroiliac Joint Pain
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Stratus Medical, INC (Unknown)
Responsible Party: Principal Investigator, Aaron Conger, Principle Investigator; Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB 150067
Record Dates: First submitted 2022-06-03; First posted 2022-06-08 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Sacroiliac Joint Complex; Low Back Pain
Keywords: Sacroiliac Joint
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: To compare pain and disability outcomes in patients with confirmed SIJC pain after randomization to either N-SIJRFA or C-SIJRFA.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to the group to which they are randomized. Given inherent approach differences between techniques, the physician performing the procedure cannot be blinded. However, staff responsible for outcome collection will remain blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nimbus Sacroiliac Joint Radiofrequency Ablation (N-SIJRFA) (Active Comparator): N-SIJRFA - using a bipolar "palisade" technique to create a continuous strip lesion.
  Interventions: Procedure: Nimbus Sacroiliac Joint Radiofrequency Ablation (N-SIJRFA)
- Conventional Sacroiliac Joint Radiofrequency Ablation (C-SIJRFA) (Active Comparator): C-SIJRFA - using conventional monopolar periforaminal technique
  Interventions: Procedure: Conventional Sacroiliac Joint Radiofrequency Ablation (C-SIJRFA)

INTERVENTIONS:
Procedure: Nimbus Sacroiliac Joint Radiofrequency Ablation (N-SIJRFA) — * Electrodes are positioned along the lateral sacral crest lateral to the inflection points of the S1, S2 and S3 lateral foraminal walls along first to third transverse sacral tubercles maintaining a craniocaudal line with an interelectrode distance of no more than 15mm.
  * The appropriate locations are confirmed in both AP and lateral views and the tines are deployed. Following injection of lidocaine, lesions are performed at 85 degrees Celsius for 180 seconds at each site for bipolar sites and 80 degrees Celsius for 90 seconds for the monopolar site. Following ablation, the tines are retracted for all electrodes prior to removal.
  Arms: Nimbus Sacroiliac Joint Radiofrequency Ablation (N-SIJRFA)
Procedure: Conventional Sacroiliac Joint Radiofrequency Ablation (C-SIJRFA) — * To target the L4 medial branch and L5 dorsal ramus, an electrode will be placed in parallel between the junction of the L5 transverse process and superior articular process and the sacral ala and S1 superior articular process.
  * A periforaminal electrode position will be used to target the lateral branches from S1 to S3. An 22-G cannula with a 5-mm exposed tip will be directed to a location approximately 3-5mm lateral to the PSFA of S1, S2, and S3. The "analog clock" positions for the probes at S1 and S2 levels will be 1:00, 3:00, and 5:30 on the right, and 6:30, 9:00, and 11:00 on the left. For the S3 level the positions at 1:30 and 4:30 on the right, and 7:30 and 10:30 on the left will be used (6,18).
  * The appropriate locations are confirmed in both AP and lateral views. Following injection of lidocaine, monopolar RFA is performed for 90 seconds at 80 degrees Celsius at each location.
  Arms: Conventional Sacroiliac Joint Radiofrequency Ablation (C-SIJRFA)

SUMMARY:
Specific Aims The sacroiliac joint complex (SIJC) is a diathrodial, synovial joint and posterior ligamentous network that receives both anterior innervation from the lumbosacral plexus as well as posterior sensory innervation via the posterior sacral network (PSN). The PSN is comprised by the lateral branches S1-S3 posterior rami, with variable contributions from S4 lateral branch, L4 medial branch, and L5 dorsal ramus. Pain signals originating from the SIJC can be interrupted with image-guided percutaneous radiofrequency ablation (RFA) of the PSN, thereby reducing pain and disability in carefully selected patients.

A prior systematic review estimated that 32-89% of patients achieve at least 50% pain relief for six months after some type of PSN ablation. Many experts suspect that heterogenous RFA techniques and technology are responsible for the variable success rates seen across published studies. Cadaveric work suggests that targeting the PSN with a large bipolar strip lesions would result in >95% PSN neural capture compared to a smaller lesion produced by a conventional, monopolar, periforaminal RFA technique which may capture as low as 2.5% of the PSN. Nimbus is a commonly used multi-tined RFA probe whose large bipolar lesion size make it an ideal option for complete PSN neural ablation. Both the Nimbus (N-SIJRFA) and conventional (C-SIJRFA) techniques and technologies are commonly used; however, there are no prospective RCT's comparing them, and the clinical significance remains unknown.

Problem: There are no randomized controlled trials comparing novel technologies like N-SIJRFA to C-SIJRFA.

Purpose: To compare pain and disability outcomes in patients with confirmed SIJC pain after randomization to either N-SIJRFA or C-SIJRFA.

Central Hypothesis: N-SIJRFA will be more effective in improving pain and function compared to patients treated with C-SIJRFA at 3, 6, 12, 18, and 24 months.

Specific Aims:

1. Compare the proportion of participants who report ≥50% relief of pain by Numeric Pain Rating Scale (NPRS) after N-SIJRFA versus C-SIJRFA.
2. Compare the proportion of participants who report ≥15-point ODI (Oswestry Disability Index) reduction after N-SIJRFA versus C-SIJRFA.
3. Compare the proportion of participants with clinically significant improvement in the categorical EuroQol 5 Dimensions tool (EQ-5D) defined by ≥0.03, after N-SIJRFA versus C-SIJRFA.
4. Compare the proportions of participants who report being "improved" or "much improved" on the Patient Global Impression of Change (PGIC) scale after N-SIJRFA versus C-SIJRFA.
5. Evaluate the differences in success rates for pain improvement, functional improvement and satisfaction in those experiencing ≥ 50%, ≥ 80%, and 100% pain relief after either prognostic PSN blocks or intra-articular (IA) sacroiliac joint (SIJ) injections.
6. Determine the effect of PSN ablation on reducing pain related sleep disturbance as measured by the Pain and Sleep Questionnaire (PSQ-3).
7. Compare procedural time requirements between those treated with N-SIJRFA versus C-SIJRFA.
8. Report adverse effects.
9. Report rates of subsequent interventional healthcare utilization including repeat N-SIJRFA versus C-SIJRFA, SIJ injection, and SIJ fusion.

DETAILED DESCRIPTION:
Low back pain affects the majority of individuals at some time in their lives. The estimated point prevalence of low back pain in 2015 was 7.3%, indicating that 540 million may be affected at any given time (1). The etiology of low back pain may be multifactorial but commonly is often attributed to nociception arising sacroiliac joint complex (SIJC) in as many as 15-30% of patients (2). The SIJC is a diathrodial, synovial joint that receives both anterior innervation from the lumbosacral plexus as well as posterior sensory innervation via the posterior sacral network (PSN) (3). The PSN is comprised by the lateral branches S1-S3 posterior rami, with variable contributions from S4 lateral branch, L4 medial branch, and L5 dorsal ramus (3-6). These have been targeted for neurotomy most commonly with image-guided percutaneous radiofrequency ablation (RFA) (7), but also with percutaneous cryoneurolysis (8), chemical neurolysis (9), endoscopic-guided RFA (10), and MRI high frequency ultrasound treatment (MRI-HIFU) (11).

Prior systematic review has suggested that 32-89% of patients may achieve at least 50% pain relief for six months, while 11-44% of patients achieved 100% pain relief for the same period (12). Although elements of patient selection likely affect this estimate (13), studies have used a variety of different RFA techniques to target the PSN which also may impact success rates. Few studies have directly compared these techniques, but cadaveric work has suggested that targeting the PSN with bipolar strip lesions results in substantially higher rates of neural capture compared to periforaminal RFA performed with conventional monopolar electrodes (6). Further, the rate of complete neural capture with a periforaminal conventional monopolar RFA may be as low as 12.5%, which is perhaps one reason why some clinical studies have shown increased probability of success in groups treated with technologies known to create larger lesions (13,14). Similar effectiveness has been observed for periforaminal techniques with both conventional monopolar compared to larger cooled monopolar lesions (15), as well as between large continuous-lesion multi-electrode lesioning compared to periforaminal conventional monopolar technique (16). However, no study has directly compared a bipolar strip lesion using a "palisade" technique (N-SIJRFA) to a conventional monopolar periforaminal method, the latter of which is used commonly in many practice settings.

The primary purpose of the current study is to evaluate the effectiveness of RFA of the PSN using a bipolar "palisade" technique to create a continuous strip lesion compared to conventional monopolar periforaminal technique in the treatment of patients with sacroiliac joint complex pain. Given the findings of recent cadaveric studies, the results of the proposed work may substantially impact the current treatment paradigm for PSN neurotomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants aged 18-90 years old with at least 3 months of low back pain who have not responded to at least 3 months of conservative treatment.
* 7-day average NPRS for low back pain of at least 4/10 at baseline
* Pain relieved by at least 50% by either a fluoroscopically-guided intraarticular sacroiliac joint injection including a local anesthetic and a fluoroscopically-guided PSN block or dual fluoroscopically-guided PSN blocks.
* Participants capable of understanding and providing consent in English and capable of complying with the outcome instruments used.

A pain diary with appropriate diagnostic categories of relief (100% relief, 80-99% relief, etc.), will be provided. Duration of pain relief will not be used as it has been shown to only marginally improve diagnostic confidence (17).

Exclusion Criteria:

* History of SIJ fusion.
* Prior SIJ RFA procedure
* Symptomatic hip osteoarthritis
* Active lumbar radicular pain
* Evidence of hardware loosening (in participants with history lumbar or lumbosacral fusion).
* Presence of pacemaker or neurostimulator.
* Chronic widespread pain or somatoform disorder (e.g., fibromyalgia).
* More than 50 mg morphine-equivalent per day opioid use.
* Active bacterial infection or treatment of infection with antibiotics within the past 4 weeks.
* Medical conditions causing significant functional disability (e.g., stroke, COPD).
* Addictive behavior, severe clinical depression, or psychotic features.
* History of anaphylactic reaction to any medication used.
* Those receiving remuneration for their pain treatment (e.g., disability, worker's compensation).
* Those involved in active litigation relevant to their pain.
* The participant is incarcerated.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Percent in NPRS Pain Score | 3 month
  The proportion of participants with ≥50% change in NPRS pain score at the 3-month follow-up assessment.

SECONDARY OUTCOMES:
Percent of Relief | 6 month
  The proportion of participants with ≥50%, relief of pain by NPRS
Percent of Relief | 12 month
  The proportion of participants with ≥50%, relief of pain by NPRS
Percent of Relief | 18 month
  The proportion of participants with ≥50%, relief of pain by NPRS
Percent of Relief | 24 month
  The proportion of participants with ≥50%, relief of pain by NPRS
ODI Reduction | 3 month
  The proportion of participants who report ≥15-point ODI reduction
ODI Reduction | 6 month
  The proportion of participants who report ≥15-point ODI reduction
ODI Reduction | 12 month
  The proportion of participants who report ≥15-point ODI reduction
ODI Reduction | 18 month
  The proportion of participants who report ≥15-point ODI reduction
ODI Reduction | 24 month
  The proportion of participants who report ≥15-point ODI reduction
EQ-5D Improvement | 3 month
  The proportion of patients with clinically significant improvement in the categorical EuroQol 5 Dimensions tool (EQ-5D) (20) defined by ≥0.03 following treatments
EQ-5D Improvement | 6 month
  The proportion of patients with clinically significant improvement in the categorical EuroQol 5 Dimensions tool (EQ-5D) (20) defined by ≥0.03 following treatments
EQ-5D Improvement | 12 month
  The proportion of patients with clinically significant improvement in the categorical EuroQol 5 Dimensions tool (EQ-5D) (20) defined by ≥0.03 following treatments
EQ-5D Improvement | 18 month
  The proportion of patients with clinically significant improvement in the categorical EuroQol 5 Dimensions tool (EQ-5D) (20) defined by ≥0.03 following treatments
EQ-5D Improvement | 24 month
  The proportion of patients with clinically significant improvement in the categorical EuroQol 5 Dimensions tool (EQ-5D) (20) defined by ≥0.03 following treatments
PGIC Improvement | 3 month
  The proportions of participants who report being "improved" or "much improved" on the Patient Global Impression of Change (PGIC) scale
PGIC Improvement | 6 month
  The proportions of participants who report being "improved" or "much improved" on the Patient Global Impression of Change (PGIC) scale
PGIC Improvement | 12 month
  The proportions of participants who report being "improved" or "much improved" on the Patient Global Impression of Change (PGIC) scale
PGIC Improvement | 18 month
  The proportions of participants who report being "improved" or "much improved" on the Patient Global Impression of Change (PGIC) scale
PGIC Improvement | 24 month
  The proportions of participants who report being "improved" or "much improved" on the Patient Global Impression of Change (PGIC) scale

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Utah Farmington Health Center, Farmington, Utah
  - University of Utah Orthopaedic Center, Salt Lake City, Utah
  - University of Utah South Jordan Health Center, South Jordan, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2015 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 310 diseases and injuries, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1545-1602. doi: 10.1016/S0140-6736(16)31678-6. PMID 27733282
- [Background] Cohen SP, Chen Y, Neufeld NJ. Sacroiliac joint pain: a comprehensive review of epidemiology, diagnosis and treatment. Expert Rev Neurother. 2013 Jan;13(1):99-116. doi: 10.1586/ern.12.148. PMID 23253394
- [Background] Roberts SL, Burnham RS, Ravichandiran K, Agur AM, Loh EY. Cadaveric study of sacroiliac joint innervation: implications for diagnostic blocks and radiofrequency ablation. Reg Anesth Pain Med. 2014 Nov-Dec;39(6):456-64. doi: 10.1097/AAP.0000000000000156. PMID 25304483
- [Background] SOLONEN KA. The sacroiliac joint in the light of anatomical, roentgenological and clinical studies. Acta Orthop Scand Suppl. 1957;27:1-127. No abstract available. PMID 13478452
- [Background] Bradley KC. The anatomy of backache. Aust N Z J Surg. 1974 Jul;44(3):227-32. doi: 10.1111/j.1445-2197.1974.tb04409.x. No abstract available. PMID 4282245
- [Background] Roberts SL, Stout A, Loh EY, Swain N, Dreyfuss P, Agur AM. Anatomical Comparison of Radiofrequency Ablation Techniques for Sacroiliac Joint Pain. Pain Med. 2018 Oct 1;19(10):1924-1943. doi: 10.1093/pm/pnx329. PMID 29415262
- [Background] Shih CL, Shen PC, Lu CC, Liu ZM, Tien YC, Huang PJ, Chou SH. A comparison of efficacy among different radiofrequency ablation techniques for the treatment of lumbar facet joint and sacroiliac joint pain: A systematic review and meta-analysis. Clin Neurol Neurosurg. 2020 Aug;195:105854. doi: 10.1016/j.clineuro.2020.105854. Epub 2020 Apr 19. PMID 32353665
- [Background] Sahoo RK, Das G, Pathak L, Dutta D, Roy C, Bhatia A. Cryoneurolysis of Innervation to Sacroiliac Joints: Technical Description and Initial Results-A Case Series. A A Pract. 2021 Mar 30;15(4):e01427. doi: 10.1213/XAA.0000000000001427. PMID 33783380
- [Background] Nouer Frederico T, Ferraro LHC, Lemos JD, Sakata RK. Chemical neurolysis of the lateral branches of the sacral dorsal rami for the treatment of chronic pain in the sacroiliac joint: Case report and description of the technique. Pain Pract. 2022 Jan;22(1):134-136. doi: 10.1111/papr.13046. Epub 2021 Jun 25. No abstract available. PMID 34077624
- [Background] Ibrahim R, Telfeian AE, Gohlke K, Decker O. Endoscopic Radiofrequency Treatment of the Sacroiliac Joint Complex for Low Back Pain: A Prospective Study with a 2-Year Follow-Up. Pain Physician. 2019 Mar;22(2):E111-E118. PMID 30921988
- [Background] Najafi A, Sartoretti E, Binkert CA. Sacroiliac Joint Ablation Using MR-HIFU. Cardiovasc Intervent Radiol. 2019 Sep;42(9):1363-1365. doi: 10.1007/s00270-019-02263-0. Epub 2019 Jun 11. PMID 31187230
- [Background] Bogduk N. Commentary on King W, Ahmed S, Baisden J, Patel N, MacVicar J, Kennedy DJ. Diagnosis of posterior sacroiliac complex pain: a systematic review with comprehensive analysis of the published data. Pain Med. 2015 Feb;16(2):222-4. doi: 10.1111/pme.12615. Epub 2014 Nov 5. No abstract available. PMID 25371349
- [Background] Cohen SP, Strassels SA, Kurihara C, Crooks MT, Erdek MA, Forsythe A, Marcuson M. Outcome predictors for sacroiliac joint (lateral branch) radiofrequency denervation. Reg Anesth Pain Med. 2009 May-Jun;34(3):206-14. doi: 10.1097/AAP.0b013e3181958f4b. PMID 19587617
- [Background] Tinnirello A, Barbieri S, Todeschini M, Marchesini M. Conventional (Simplicity III) and Cooled (SInergy) Radiofrequency for Sacroiliac Joint Denervation: One-Year Retrospective Study Comparing Two Devices. Pain Med. 2017 Sep 1;18(9):1731-1744. doi: 10.1093/pm/pnw333. PMID 28340063
- [Background] Cheng J, Pope JE, Dalton JE, Cheng O, Bensitel A. Comparative outcomes of cooled versus traditional radiofrequency ablation of the lateral branches for sacroiliac joint pain. Clin J Pain. 2013 Feb;29(2):132-7. doi: 10.1097/AJP.0b013e3182490a17. PMID 22688606
- [Background] Speldewinde GC. Successful Thermal Neurotomy of the Painful Sacroiliac Ligament/Joint Complex-A Comparison of Two Techniques. Pain Med. 2020 Mar 1;21(3):561-569. doi: 10.1093/pm/pnz282. PMID 31747020
- [Background] Bogduk N. On the Rational Use of Diagnostic Blocks for Spinal Pain. Neurosurg Q. 2009 Jun;19(2):88-100.
- [Background] Cohen SP, Hurley RW, Buckenmaier CC 3rd, Kurihara C, Morlando B, Dragovich A. Randomized placebo-controlled study evaluating lateral branch radiofrequency denervation for sacroiliac joint pain. Anesthesiology. 2008 Aug;109(2):279-88. doi: 10.1097/ALN.0b013e31817f4c7c. PMID 18648237
- [Background] Copay AG, Glassman SD, Subach BR, Berven S, Schuler TC, Carreon LY. Minimum clinically important difference in lumbar spine surgery patients: a choice of methods using the Oswestry Disability Index, Medical Outcomes Study questionnaire Short Form 36, and pain scales. Spine J. 2008 Nov-Dec;8(6):968-74. doi: 10.1016/j.spinee.2007.11.006. Epub 2008 Jan 16. PMID 18201937
- [Background] Soer R, Reneman MF, Speijer BL, Coppes MH, Vroomen PC. Clinimetric properties of the EuroQol-5D in patients with chronic low back pain. Spine J. 2012 Nov;12(11):1035-9. doi: 10.1016/j.spinee.2012.10.030. PMID 23199409
- [Background] Ayearst L, Harsanyi Z, Michalko KJ. The Pain and Sleep Questionnaire three-item index (PSQ-3): a reliable and valid measure of the impact of pain on sleep in chronic nonmalignant pain of various etiologies. Pain Res Manag. 2012 Jul-Aug;17(4):281-90. doi: 10.1155/2012/635967. PMID 22891194
- [Background] Tonosu J, Oka H, Watanabe K, Abe H, Higashikawa A, Kawai T, Yamada K, Nakarai H, Tanaka S, Matsudaira K. Characteristics of the spinopelvic parameters of patients with sacroiliac joint pain. Sci Rep. 2021 Mar 4;11(1):5189. doi: 10.1038/s41598-021-84737-1. PMID 33664386
- [Background] Tonosu J, Kurosawa D, Nishi T, Ito K, Morimoto D, Musha Y, Ozawa H, Murakami E. The association between sacroiliac joint-related pain following lumbar spine surgery and spinopelvic parameters: a prospective multicenter study. Eur Spine J. 2019 Jul;28(7):1603-1609. doi: 10.1007/s00586-019-05952-z. Epub 2019 Mar 18. PMID 30887220